CLINICAL TRIAL: NCT00569452
Title: Comparison of Basal (Fasting) Glycemic Control in Type 1 Diabetic Patients With CSII Achieved by the Circadian Slide Ruler Scale or Flat Basal Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000278; DMS-01-CIRCADIAN-01
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- A (Experimental)
  Interventions: Device: Accu-Chek Spirit Insulin Pump
- B (Experimental)
  Interventions: Device: Accu-Chek Spirit Insulin Pump

INTERVENTIONS:
Device: Accu-Chek Spirit Insulin Pump — One basal rate
  Arms: A
Device: Accu-Chek Spirit Insulin Pump — Multiple basal rates
  Arms: B

SUMMARY:
This is a pilot trial to establish study procedures that allow comparison of various starting basal rate profiles used in Continuous Subcutaneous Insulin Infusion (CSII). Glycemic control achieved by circadian 'slide ruler scale' basal rate versus that achieved by one constant basal rate (flat profile) will be compared during a composite fasting day as well as therapeutic success after 2 weeks of normal activity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years of age
* Type 1 diabetes
* Diabetic for >2 years, and treated with CSII for >= 3 months
* HbA1c <=8.5%

Exclusion Criteria:

* Excessive fibrosis or lipo-hypertrophy at injection or infusion sites
* Unstable chronic disease other than type 1 diabetes
* Severe hypoglycemic event within last week prior to study start
* Severe diabetic ketoacidosis within last month prior to study start

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Pilot trial to establish endpoints such as "time within target range of a composite fasting day" | Study duration

SECONDARY OUTCOMES:
AUC, MAGE, HbA1c, body weight change | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Buhr, Study Director — Disetronic Medical Systems AG
Locations (1):
- Ulm, Germany